CLINICAL TRIAL: NCT02845895
Title: Study to Compare Strategies to Improve Detection of Nutritional Disorders in Hospitalized Adults (Compass Project)
Acronym: CompaS
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 12 557 15
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Nutritional Disorder
Keywords: Screening for nutritional disorder; Comparison of two organizations; Indicator IPAQSS
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neuroscience pole: Patient hospitalized in the department of medicine-surgery-obstetric of the neuroscience pole department
  Interventions: Other: Caregiver dedicated
- Respiratory tracts pole: Patient hospitalized in the department of medicine-surgery-obstetric of the respiratory tracts pole department
  Interventions: Other: Classic strategy

INTERVENTIONS:
Other: Caregiver dedicated — Organization of nutrition screening with the help of a caregiver
  Groups: Neuroscience pole
Other: Classic strategy — Classic organization with the training of the department team
  Groups: Respiratory tracts pole

SUMMARY:
The prevalence of malnutrition in hospital is very high (30 percent) with major consequences in terms of morbidity and mortality, generating significant health care costs. The positive impact of its support is demonstrated.

The HAS (French High Sanitary Authority) recommends a screening of all adult hospitalized in the first 48 hours, with no consensus regarding the organization of screening within care services. Various strategies have been implemented. Although this screening is part of the nursing role, old and recent studies show that it is not done systematically and nutritional disorders are largely under-diagnosed and therefore untreated.

The investigators assume that an organization of screening for eating disorders, based on a caregiver dedicated to this activity, improves the indicator IPAQSS (Indicateurs Pour l'Amélioration de la Qualité et de la Sécurité des Soins) which is an indicator for the improvement of the quality and security of care) Screening indicator of nutritional disorders Level 3, compared to an organization "classic" involving the care teams in their entirety. This indicator reflects the care system performance.

In this study, patients will have no intervention. Only the organization of the care staff will be adapted but with no changes on the care of patients?

DETAILED DESCRIPTION:
Undernutrition in the hospital is a public health issue. The impacts of this malnutrition are known , with consequences clearly established on the morbidity, mortality and quality of life. Undernutrition is an independent risk factor for mortality (5). In terms of morbidity, the most frequently reported consequences are infections, postoperative complications (delayed healing, in particular nosocomial infections, risk of pressure ulcers) and pejorative impact on the prognosis of chronic diseases such as respiratory failure , heart and kidney.

Malnutrition therefore affects the length of hospital stays and the burden of care.

Many studies have shown the positive impact of the medical care of malnutrition on morbidity and mortality, whether intervention studies in general hospital population or in specific pathologies.

But there is no systematic screening strategy undernutrition implementation in hospitals.

The investigators assume that the organization of screening for eating disorders based on a caregiver specifically dedicated to this activity, improves the indicator IPAQSS Screening indicator of nutritional disorders level 3 compared with a "classic" organization shared between different actors of care. This indicator reflects the care system performance This organization must advance quickly and significantly the number of patients evaluated nutritionally and help reach a level of completeness close to 100%.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in medicine-surgery-obstetrics department
* Patient over 18 years

Exclusion Criteria:

* Patient hospitalized less than 48 hours
* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the department of medicine-surgery-obstetric
Sampling Method: Non-Probability Sample
Enrollment: 916 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change of patients responding at the level 3 of IPAQSS criterion | Before the surgery and 6 months after the surgery

SECONDARY OUTCOMES:
Change of patients responding at the level 2 of IPAQSS criterion | Before the surgery and 6 months after the surgery
Change of the cost-efficiency | Before the surgery and 6 months after the surgery
  The cost of hospitalization between the 2 arms will be compared
Change of patients responding at the level 3 and level 2 of IPAQSS criterion | 15 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Monelle Bertrand, MD, PhD, Principal Investigator — Hospital University of Toulouse
Locations (1):
- Centre hospitalier Universitaire de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schindler K, Pernicka E, Laviano A, Howard P, Schutz T, Bauer P, Grecu I, Jonkers C, Kondrup J, Ljungqvist O, Mouhieddine M, Pichard C, Singer P, Schneider S, Schuh C, Hiesmayr M; NutritionDay Audit Team. How nutritional risk is assessed and managed in European hospitals: a survey of 21,007 patients findings from the 2007-2008 cross-sectional nutritionDay survey. Clin Nutr. 2010 Oct;29(5):552-9. doi: 10.1016/j.clnu.2010.04.001. PMID 20434820
- [Background] Imoberdorf R, Meier R, Krebs P, Hangartner PJ, Hess B, Staubli M, Wegmann D, Ruhlin M, Ballmer PE. Prevalence of undernutrition on admission to Swiss hospitals. Clin Nutr. 2010 Feb;29(1):38-41. doi: 10.1016/j.clnu.2009.06.005. Epub 2009 Jul 1. PMID 19573958
- [Background] Korfali G, Gundogdu H, Aydintug S, Bahar M, Besler T, Moral AR, Oguz M, Sakarya M, Uyar M, Kilicturgay S. Nutritional risk of hospitalized patients in Turkey. Clin Nutr. 2009 Oct;28(5):533-7. doi: 10.1016/j.clnu.2009.04.015. Epub 2009 May 28. PMID 19481309
- [Background] Sorensen J, Kondrup J, Prokopowicz J, Schiesser M, Krahenbuhl L, Meier R, Liberda M; EuroOOPS study group. EuroOOPS: an international, multicentre study to implement nutritional risk screening and evaluate clinical outcome. Clin Nutr. 2008 Jun;27(3):340-9. doi: 10.1016/j.clnu.2008.03.012. Epub 2008 May 27. PMID 18504063
- [Background] Correia MI, Waitzberg DL. The impact of malnutrition on morbidity, mortality, length of hospital stay and costs evaluated through a multivariate model analysis. Clin Nutr. 2003 Jun;22(3):235-9. doi: 10.1016/s0261-5614(02)00215-7. PMID 12765661
- [Background] Norman K, Pichard C, Lochs H, Pirlich M. Prognostic impact of disease-related malnutrition. Clin Nutr. 2008 Feb;27(1):5-15. doi: 10.1016/j.clnu.2007.10.007. Epub 2007 Dec 3. PMID 18061312
- [Background] Lim SL, Daniels L. Reply--Malnutrition and its impact on cost of hospitalization, length of stay, readmission and 3-year mortality. Clin Nutr. 2013 Jun;32(3):489-90. doi: 10.1016/j.clnu.2012.12.014. Epub 2013 Jan 11. No abstract available. PMID 23347962
- [Background] Starke J, Schneider H, Alteheld B, Stehle P, Meier R. Short-term individual nutritional care as part of routine clinical setting improves outcome and quality of life in malnourished medical patients. Clin Nutr. 2011 Apr;30(2):194-201. doi: 10.1016/j.clnu.2010.07.021. PMID 20937544
- [Background] Johansen N, Kondrup J, Plum LM, Bak L, Norregaard P, Bunch E, Baernthsen H, Andersen JR, Larsen IH, Martinsen A. Effect of nutritional support on clinical outcome in patients at nutritional risk. Clin Nutr. 2004 Aug;23(4):539-50. doi: 10.1016/j.clnu.2003.10.008. PMID 15297090
- [Background] Norman K, Kirchner H, Freudenreich M, Ockenga J, Lochs H, Pirlich M. Three month intervention with protein and energy rich supplements improve muscle function and quality of life in malnourished patients with non-neoplastic gastrointestinal disease--a randomized controlled trial. Clin Nutr. 2008 Feb;27(1):48-56. doi: 10.1016/j.clnu.2007.08.011. Epub 2007 Oct 25. PMID 17964008
- [Background] Braga M, Gianotti L, Vignali A, Carlo VD. Preoperative oral arginine and n-3 fatty acid supplementation improves the immunometabolic host response and outcome after colorectal resection for cancer. Surgery. 2002 Nov;132(5):805-14. doi: 10.1067/msy.2002.128350. PMID 12464864
- [Background] Kruizenga HM, Van Tulder MW, Seidell JC, Thijs A, Ader HJ, Van Bokhorst-de van der Schueren MA. Effectiveness and cost-effectiveness of early screening and treatment of malnourished patients. Am J Clin Nutr. 2005 Nov;82(5):1082-9. doi: 10.1093/ajcn/82.5.1082. PMID 16280442
- [Background] Elia M, Zellipour L, Stratton RJ. To screen or not to screen for adult malnutrition? Clin Nutr. 2005 Dec;24(6):867-84. doi: 10.1016/j.clnu.2005.03.004. PMID 15893857